CLINICAL TRIAL: NCT05157425
Title: Efficacy and Safety of a Multistrain Probiotic Formula to Boost the Immune Response to Influenza Virus Vaccination
Brief Title: Effect of a Multi-strain Probiotic Formulation on Immune Response to Influenza Vaccination
Acronym: FLUVAC21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AB-FLUVAC21
Record Dates: First submitted 2021-11-19; First posted 2021-12-15 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Influenza Vaccine
Keywords: influenza vaccination, probiotic
MeSH Terms: conditions — Influenza, Human | interventions — Dietary Supplements; Probiotics

STUDY DESIGN:
Intervention Model Description: Double blind, randomized controlled trial in 140 subjects 50-80 years old receiving influenza vaccination, who will be allocated to receive either an experimental product containing multi-strain probiotic formula or placebo for 28 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both placebo and active product will be provided in identical packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Probiotic multi-strain formulation comprising L. plantarum CECT30292, CECT7484, CECT7585 and P. acidilactici and maltodextrin (E1400, qs) as excipient in hydroxymethylpropyl-cellulose (HPMC) capsules. Probiotic strains have Qualified Presumption of Safety (QPS) status by European Food Safety Authority
  Interventions: Dietary Supplement: Food Supplement
- Placebo (Placebo Comparator): Maltodextrin (E1400, qs) in HPMC capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food Supplement — Probiotic multistrain formulation containing Lactiplantibacillus plantarum CECT30292, CECT7484, CECT7485 and P. acidilactici CECT7483 for 28 days, starting the same day of influenza vaccination
  Other Names: Probiotic
  Arms: Experimental
Dietary Supplement: Placebo — One maltodextrin-containing capsule/day for 28 days, starting the same day of influenza vaccination
  Arms: Placebo

SUMMARY:
Randomized clinical trial to determine whether a probiotic formulation containing 4 probiotic strains which belong to Lactiplantibacillus plantarum and Pediococcus acidilactici species can boost the immune response to influenza vaccination evaluated at 4 weeks in a population between 50 and 80 years of age. Secondary outcomes comprise evaluation of immune response at 8 weeks after vaccination, percentage of patients with seroconversion, incidence and duration of influenza-like infections and respiratory infections throughout a 4-month period and safety.

DETAILED DESCRIPTION:
Double blind, randomized, placebo-controlled clinical trial to determine whether supplementation with a probiotic formulation containing 4 probiotic strains (L. plantarum CECT 30292, CECT7484, CECT7485 and P. acidilactici CECT7483) can improve immune response to seasonal influenza vaccination. Subjects with age comprised between 50 and 80 years who meet inclusion and exclusion criteria will be randomized 1:1 to one of the following study groups: one will receive probiotic formulation for 28 days (1 capsule/day) and the other will receive placebo, starting the same day of the influenza vaccination. Main study outcome will be immune response at 4 weeks after vaccination, which will be determined by analysis of specific IgG antibodies in serum against influenza A and B. Secondary outcomes comprise serum titers of specific IgG at 8 weeks after vaccination, percentage of patients with seroconversion at 4 and 8 weeks, evaluation of influenza-like infections or respiratory infections throughout a 4-month period and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 50 - 80 years old receiving seasonal Influenza vaccine in season 2021-2022
* Body mass index (BMI) 18.5-34.9 kg/m2
* Willing to provide informed consent
* Able to follow study procedures, according to the criteria of study investigator

Exclusion Criteria:

* Hypersensitivity to any of the components of influenza vaccine
* Previous influenza infection in the same season (from 01/09/2021)
* Having received influenza vaccination in the previous season less than 9 months before study entry (from 01/01/2021)
* Having received another vaccine -different from COVID19 vaccine- up to 1 month before study inclusion or planning to receive it 1 month after study inclusion
* Active infection at the moment of study entry as diagnosed by study physician
* History of severe allergic reactions (food and non-food), including severe asthma.
* Receiving immunosuppressant therapy, displaying neutropenia, lymphopenia, AIDS, immunoglobulin deficiency, active oncological disease.
* Daily ingestion of any food complement or food added with probiotics (including Actimel o similar products) 2 weeks before inclusion in the study
* Acute pancreatitis, short bowel syndrome or active inflammatory bowel disease
* Diagnosed from other pathologies that according to study physician may compromise the immunological function of the individual (such as immunodeficiencies, lupus, multiple sclerosis, among others)
* Having received antibiotic treatment in the previous month

Exclusion criteria during the study:

* Withdrawal from the study as per study investigator criteria, in case that study procedures are not followed by the participant
* In case of adverse event that prevents them from following study procedures or complying with the treatments under study.
* Failure to comply with study procedures: Complete less than 70% of the days in the patient's diary and/or take less than 80% of the days of the study products.
* Receive any of the unauthorized treatments indicated in the selection criteria, with the exception of antibiotics that will be allowed under medical prescription.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
IgG antibodies against vaccine influenza antigens | 4 weeks (day 1 and day 28)
  Titer of specific total IgG antibodies against vaccine influenza A and B antigens at day 28

SECONDARY OUTCOMES:
IgG antibodies against vaccine influenza antigens | 8 weeks (day 1 and day 56)
  Titer of specific total IgG antibodies against vaccine influenza A and B antigens at day 56
IgM antibodies against vaccine influenza antigens | 8 weeks (day 1 and day 56)
  Titer of specific total IgM antibodies against vaccine influenza A and B antigens at day 28 and 56
Seroconversion | 8 weeks (day 1,day 28 and 56)
  Percentage of patients with seroconversion (defined as 4 fold change in influenza IgG antibodies concentration compared to baseline) at day 28 and 56
Incidence of influenza like infections (ILI) | 16 weeks (day 1, day 56)
  Cumulative incidence of influenza like infection (ILI), according to the European Diseases Prevention and Control Center (ECDC) criteria
Incidence of any other respiratory infections (including COVID-19) | 16 weeks (day 1, day 56)
  Cumulative incidence of any other respiratory infections
Incidence of fever | 16 weeks (day 1, day 56)
  Cumulative number of days with fever (> 37.5ºC)
Use of analgesics and antibiotics | 16 weeks (day 1, day 56)
  Cumulative number of days using analgesics and antibiotics
Duration of vaccine-related symptoms: injection-site pain, swelling, redness | 1 week (day 1, day 7)
  Duration (in days) of symptoms after receiving the flu vaccine.
Severity of vaccine-related symptoms: injection-site pain, swelling, redness | 1 week (day 1, day 7)
  Severity of symptoms after receiving the flu vaccine. Measured on a 4-point scale: 0 = none , 1 = mild, 2 = moderate, and 3 = severe
Gastrointestinal symptoms | 4 weeks (day 1, day 28)
  Gastrointestinal manifestations documented through questionnaire in participants diary. Measured on a 4-point scale: 0 = none , 1 = mild, 2 = moderate, and 3 = severe.
Adverse events | 8 weeks (day 56)
  Frequency of adverse events reported in medical visits or patient diary
Albumin | 4 weeks (day 1, day 28)
  Albumin concentration in blood
Alkaline phosphatase (ALP) | 4 weeks (day 1, day 28)
  Alkaline phosphatase (ALP) concentration in blood
Gamma-glutamil transpeptidase (GGT) | 4 weeks (day 1, day 28)
  Gamma-glutamil transpeptidase (GGT) concentration in blood
Aspartate aminotransferase (GOT) | 4 weeks (day 1, day 28)
  Aspartate aminotransferase (AST) concentration in blood
Alanine aminotransferase (AST) | 4 weeks (day 1, day 28)
  Aspartate aminotransferase (AST) concentration in blood
Basic hemogram | 4 weeks (day 1, day 28)
  Blood cell count

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Parc Tauli, Sabadell, Barcelona
  - IDIAP Jordi Gol-Centro de Atención Primaria La Mina, Sant Adrià de Besòs, Barcelona
  - Mutua de Terrassa, Terrassa, Barcelona
  - FIBAO- Fundación para la Investigación Biosanitaria de Andalucia Oriental, Granada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambert ND, Ovsyannikova IG, Pankratz VS, Jacobson RM, Poland GA. Understanding the immune response to seasonal influenza vaccination in older adults: a systems biology approach. Expert Rev Vaccines. 2012 Aug;11(8):985-94. doi: 10.1586/erv.12.61. PMID 23002979
- [Background] Ng TWY, Cowling BJ, Gao HZ, Thompson MG. Comparative Immunogenicity of Enhanced Seasonal Influenza Vaccines in Older Adults: A Systematic Review and Meta-analysis. J Infect Dis. 2019 Apr 19;219(10):1525-1535. doi: 10.1093/infdis/jiy720. PMID 30551178
- [Background] Harper A, Vijayakumar V, Ouwehand AC, Ter Haar J, Obis D, Espadaler J, Binda S, Desiraju S, Day R. Viral Infections, the Microbiome, and Probiotics. Front Cell Infect Microbiol. 2021 Feb 12;10:596166. doi: 10.3389/fcimb.2020.596166. eCollection 2020. PMID 33643929
- [Background] Trombetta CM, Remarque EJ, Mortier D, Montomoli E. Comparison of hemagglutination inhibition, single radial hemolysis, virus neutralization assays, and ELISA to detect antibody levels against seasonal influenza viruses. Influenza Other Respir Viruses. 2018 Nov;12(6):675-686. doi: 10.1111/irv.12591. Epub 2018 Aug 11. PMID 30019448
- [Background] Lynn DJ, Benson SC, Lynn MA, Pulendran B. Modulation of immune responses to vaccination by the microbiota: implications and potential mechanisms. Nat Rev Immunol. 2022 Jan;22(1):33-46. doi: 10.1038/s41577-021-00554-7. Epub 2021 May 17. PMID 34002068
- [Result] Zimmermann P, Curtis N. The influence of probiotics on vaccine responses - A systematic review. Vaccine. 2018 Jan 4;36(2):207-213. doi: 10.1016/j.vaccine.2017.08.069. Epub 2017 Sep 18. PMID 28923425
- [Result] Yeh TL, Shih PC, Liu SJ, Lin CH, Liu JM, Lei WT, Lin CY. The influence of prebiotic or probiotic supplementation on antibody titers after influenza vaccination: a systematic review and meta-analysis of randomized controlled trials. Drug Des Devel Ther. 2018 Jan 25;12:217-230. doi: 10.2147/DDDT.S155110. eCollection 2018. PMID 29416317
- [Result] Darbandi A, Asadi A, Ghanavati R, Afifirad R, Darb Emamie A, Kakanj M, Talebi M. The effect of probiotics on respiratory tract infection with special emphasis on COVID-19: Systemic review 2010-20. Int J Infect Dis. 2021 Apr;105:91-104. doi: 10.1016/j.ijid.2021.02.011. Epub 2021 Feb 9. PMID 33578007